CLINICAL TRIAL: NCT05412004
Title: A Master Protocol to Investigate the Efficacy and Safety of Tirzepatide Once Weekly in Participants Who Have Obstructive Sleep Apnea and Obesity: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Obstructive Sleep Apnea Master Protocol GPIF: A Study of Tirzepatide (LY3298176) in Participants With Obstructive Sleep Apnea
Acronym: SURMOUNT-OSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18357; I8F-MC-GPIF (Other: Eli Lilly and Company); I8F-MC-GPI1 (Other: Eli Lilly and Company); I8F-MC-GPI2 (Other: Eli Lilly and Company); 2021-004552-41 (EudraCT Number)
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tirzepatide MTD_GPI1 (Experimental): Participants not on positive airway pressure (PAP) therapy received a maximum tolerated dose (MTD) of 10 milligrams (mg) or 15 mg of Tirzepatide once weekly (QW) as a subcutaneous (SC) injection for 52 weeks, including the initial dose escalation by 2.5 mg every 4 weeks
  Interventions: Drug: Tirzepatide
- Placebo_GPI1 (Placebo Comparator): Participants not on PAP therapy received placebo QW as an SC injection for 52 weeks.
  Interventions: Drug: Placebo
- Tirzepatide MTD_GPI2 (Experimental): Participants who are on PAP therapy received an MTD of 10 mg or 15 mg of Tirzepatide QW as an SC injection for 52 weeks, including the initial dose escalation by 2.5 mg every 4 weeks
  Interventions: Drug: Tirzepatide
- Placebo_GPI2 (Placebo Comparator): Participants who are on PAP therapy received placebo QW as an SC injection for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide MTD_GPI1; Tirzepatide MTD_GPI2
Drug: Placebo — Administered SC
  Arms: Placebo_GPI1; Placebo_GPI2

SUMMARY:
The purpose of this study is to evaluate the effect and safety of tirzepatide in participants with moderate to severe obstructive sleep apnea and obesity who are both unwilling or unable to use Positive Airway Pressure (PAP) therapy in GPI1 and those who are and plan to stay on PAP therapy in GPI2.

ELIGIBILITY:
Inclusion Criteria:

For GPI1 Participants:

- Participants who are unable or unwilling to use PAP therapy. Participants must not have used PAP for at least 4 weeks prior to screening.

For GPI2 Participants:

- Have been on PAP therapy for at least 3 consecutive months prior to screening and plan to continue PAP therapy during the study

For Both GPI1 and GPI2 Participants:

* Have an AHI ≥15 on PSG as part of the trial at screening
* Have a body mass index (BMI) ≥30 kilogram/square meter (kg/m²)
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight

Exclusion Criteria:

For GPI2 Participants:

* Have personal or job-related responsibilities, or in the opinion of the investigator have any situation, that would make it unsafe to stop PAP therapy for 7 days prior to PSG testing during the course of the study
* Are unwilling to stop PAP therapy for 7 days prior to polysomnography (PSG) testing during the course of the study

For GPI1 and GPI2 Participants:

* Female participants must not be pregnant, intending to be pregnant, breastfeeding, or intending to breastfeed.
* Have type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM), history of ketoacidosis, or hyperosmolar state/coma.
* Have HbA1c ≥ 6.5% (≥ 48 mmol/mol) at baseline
* Any previous or planned surgery for sleep apnea or major ear, nose or throat surgery, including tonsillectomy and adenoidectomy that still may affect breathing at time of baseline
* Have significant craniofacial abnormalities that may affect breathing at baseline
* Have diagnosis of Central or Mixed Sleep Apnea with % of mixed or central apneas/hypopneas ≥50%, or diagnosis of Cheyne Stokes Respiration
* Diagnosis of Obesity Hypoventilation Syndrome or daytime hypercapnia.
* Active device treatment of OSA other than PAP therapy (for example, dental appliance), or other treatment, that in the opinion of the investigator, may interfere with study outcomes, unless willing to stop treatment at baseline and throughout the study.
* Respiratory and neuromuscular diseases that could interfere with the results of the trial in the opinion of the investigator.
* Have a self-reported change in body weight >5 kg within 3 months prior to screening
* Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty if performed more than 1 year prior to screening)
* Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months (for example, mucosal ablation, gastric artery embolization, intragastric balloon, and duodenal-jejunal bypass sleeve)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (57):
- United States (18):
  - Artemis Institute for Clinical Research, Riverside, California
  - Teradan Clinical Trials, LLC, Brandon, Florida
  - Renstar Medical Research, Ocala, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Brengle Family Medicine, Indianapolis, Indiana
  - Lillestol Research, Fargo, North Dakota
  - NeuroScience Research Center, Canton, Ohio
  - CTI-CRC, Cincinnati, Ohio
  - Office 18, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - Advanced Neuro Research Center - ANRC, El Paso, Texas
  - Epic Medical Research, Red Oak, Texas
  - Sleep Therapy Research Center, San Antonio, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Australia (2):
  - Woolcock Institute of Medical Research, Sydney, New South Wales
  - Flinders University, Bedford Park, South Australia
- Brazil (5):
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - CPCLIN, São Paulo, São Paulo
  - CPQuali Pesquisa Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo
- China (6):
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Praglandia s.r.o, Prague
- Germany (7):
  - Siteworks GmbH, Hanover, Lower Saxony
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Institut für Diabetesforschung GmbH Münster, Münster, North Rhine-Westphalia
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Lungenpraxis Schleswig, Schleswig, Schleswig-Holstein
  - Advanced Sleep Research, Berlin
  - Diabeteszentrum Hamburg West, Hamburg
- Japan (6):
  - Koujunkai Daido Clinic, Nagoya, Aichi-ken
  - Kirigaokatsuda Hospital, Kitakyushu, Fukuoka
  - RESM Respiratory and Sleep Medical Care Clinic, Yokohama, Kanagawa
  - Sakai City Medical Center, Sakai, Osaka
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Osaka Kaisei Hospital, Osaka
- Mexico (8):
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara, Jalisco
  - Unidad de Investigación Clínica y Atención Médica HEPA, Guadalajara, Jalisco
  - RM Pharma Specialists, Mexico City, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - Servicios Integrales Nova de Monterrey S.A. de C.V., San Nicolás de los Garza, Nuevo León
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
  - Arké SMO S.A de C.V, Veracruz
- Puerto Rico Medical Research Center, Hato Rey, Puerto Rico, Puerto Rico
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Malhotra A, Grunstein R, Azarbarzin A, Sands S, Somers VK, Aronne LJ, Jastreboff AM, Lou J, Chakladar S, Dunn JP, Bunck MC, Bednarik J. Tirzepatide on obstructive sleep apnea-related cardiometabolic risk: secondary outcomes of the SURMOUNT-OSA randomized trial. Nat Med. 2026 Jan 15. doi: 10.1038/s41591-025-04071-1. Online ahead of print. PMID 41540105
- [Derived] Malhotra A, Grunstein RR, Azarbarzin A, Sands SA, Dang X, Chakladar S, Dunn JP, Falcon B, Bednarik J. Tirzepatide for sleep-disordered breathing in SURMOUNT-OSA: Time course and association with body weight. Sleep Med. 2025 Dec;136:106853. doi: 10.1016/j.sleep.2025.106853. Epub 2025 Oct 14. PMID 41135142
- [Derived] Kanu C, Shinde S, Chakladar S, Dennehy EB, Weaver TE, Poon JL, Malhotra A. Effect of tirzepatide treatment on patient-reported outcomes among SURMOUNT-OSA participants with obstructive sleep apnea and obesity. Sleep Med. 2025 Oct;134:106719. doi: 10.1016/j.sleep.2025.106719. Epub 2025 Aug 6. PMID 40774158
- [Derived] Malhotra A, Grunstein RR, Fietze I, Weaver TE, Redline S, Azarbarzin A, Sands SA, Schwab RJ, Dunn JP, Chakladar S, Bunck MC, Bednarik J; SURMOUNT-OSA Investigators. Tirzepatide for the Treatment of Obstructive Sleep Apnea and Obesity. N Engl J Med. 2024 Oct 3;391(13):1193-1205. doi: 10.1056/NEJMoa2404881. Epub 2024 Jun 21. PMID 38912654
- [Derived] Malhotra A, Bednarik J, Chakladar S, Dunn JP, Weaver T, Grunstein R, Fietze I, Redline S, Azarbarzin A, Sands SA, Schwab RJ, Bunck MC. Tirzepatide for the treatment of obstructive sleep apnea: Rationale, design, and sample baseline characteristics of the SURMOUNT -OSA phase 3 trial. Contemp Clin Trials. 2024 Jun;141:107516. doi: 10.1016/j.cct.2024.107516. Epub 2024 Mar 26. PMID 38547961
- See also: Obstructive Sleep Apnea Master Protocol GPIF: A Study of Tirzepatide (LY3298176) in Participants With Obstructive Sleep Apnea (SURMOUNT-OSA) — https://clinicaltrials.gov/study/NCT05412004?tab=results

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NCT05412004 supports two pivotal studies: I8F-MC-GPI1 (GPI1; Study 1) and I8F-MC-GPI2 (GPI2; Study 2), conducted under the single master protocol I8F-MC-GPIF. The studies were conducted under a single overarching trial structure for operational efficiencies, but the study participants for both studies are different (GPI1 included participants who were unable or unwilling to use positive airway pressure (PAP) therapy, while GPI2 included those on PAP therapy).
Period: Overall Study
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Started | 114 | 120 | 120 | 115
Received at Least One Dose of Study Drug | 114 | 120 | 119 | 114
Completed | 101 | 86 | 113 | 89
Not Completed | 13 | 34 | 7 | 26
Not completed — Adverse Event | 0 | 2 | 1 | 5
Not completed — Assigned Treatment by Mistake | 5 | 10 | 2 | 5
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Patient could not travel to site | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 19 | 4 | 14
Not completed — Screen Failure | 0 | 0 | 0 | 1
Not completed — The participant quit treatment and study due to their schedule and the final V801 was done remotely | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2 | Total
Number analyzed (Participants) | 114 | 120 | 120 | 115 | 469
Age, Customized [Count of Participants; unit: Participants]
  <50years | 63 | 62 | 54 | 45 | 224
  >=50years | 51 | 58 | 66 | 70 | 245
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 33 | 32 | 142
  Male | 78 | 79 | 87 | 83 | 327
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 47 | 38 | 38 | 174
  Not Hispanic or Latino | 63 | 69 | 82 | 76 | 290
  Unknown or Not Reported | 0 | 4 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 9 | 10 | 9 | 37
  Asian | 23 | 24 | 17 | 16 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 8 | 3 | 24
  White | 74 | 80 | 85 | 86 | 325
  More than one race | 2 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 36 | 41 | 37 | 149
  China | 14 | 14 | 4 | 5 | 37
  Japan | 3 | 4 | 7 | 6 | 20
  Taiwan | 5 | 4 | 4 | 3 | 16
  Brazil | 24 | 25 | 18 | 17 | 84
  Mexico | 20 | 19 | 14 | 16 | 69
  Australia | 1 | 5 | 10 | 9 | 25
  Germany | 7 | 7 | 16 | 16 | 46
  Czechia | 5 | 6 | 6 | 6 | 23
Baseline apnea-hypopnea index (AHI) [Mean (Standard Deviation); unit: events per hour] — AHI is the number of apneas or hypopneas recorded via polysomnography during the study per hour of sleep. Apnea is defined as a cessation of airflow lasting at least 10 seconds, hypopnea as a decrease in airflow by at least 30% from baseline for at least 10 seconds occurring with a drop in oxygen saturation (SpO₂) by at least 4%. AHI values are categorized as 5-15 episodes/hr = mild; 15-<30 episodes/hr = moderate; and ≥ 30 episodes/h = severe. a significant reduction in values indicates a positive outcome. Population: All randomized participants. Number analysed includes subjects with non-missing data.
  events per hour
    number analyzed (Participants) | 114 | 119 | 119 | 114 | 466
    (all) | 52.86 (30.50) | 50.13 (31.47) | 46.08 (22.35) | 53.10 (30.23) | 50.49 (28.98)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Apnea-Hypopnea Index (AHI)
Description: AHI, Apnea-Hypopnea Index, is the number of apneas or hypopneas recorded via polysomnography during the study per hour of sleep. Apnea is defined as a cessation of airflow lasting at least 10 seconds, hypopnea as a decrease in airflow by at least 30% from baseline for at least 10 seconds occurring with a drop in oxygen saturation (SpO₂) by at least 4%. AHI values are categorized as 5-15 events/hr = mild; 15-<30 events/hr = moderate; and ≥ 30 events/hr = severe. a significant reduction in values indicates a positive outcome.
Time Frame: Baseline, Week 52
Population: Modified intent-to-treat (mITT) population consisting of all randomized participants who are exposed to at least 1 dose of study intervention and have evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: events per hour
Groups:
- Tirzepatide MTD_GPI1: Participants not on PAP therapy received an MTD of 10 mg or 15 mg of Tirzepatide QW as an SC injection for 52 weeks, including the initial dose escalation by 2.5 mg every 4 weeks.
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 100 | 86 | 110 | 87
events per hour | -25.25 (2.06) | -5.25 (2.11) | -29.27 (1.99) | -5.51 (2.21)
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model was used with baseline, geographic region, sex, treatment (Type III sum of squares) as covariates; LS Mean Change difference = -20.01, 95% CI 2-sided [-25.82 to -14.20]
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model was used with baseline, geographic region, sex, treatment (Type III sum of squares) as covariates; LS Mean Change difference = -23.77, 95% CI 2-sided [-29.61 to -17.93]

2. Secondary Outcome: Percent Change From Baseline in Apnea-Hypopnea Index (AHI)
Description: Percent Change From Baseline in AHI was evaluated.
Time Frame: Baseline, Week 52
Population: mITT population consisting of all randomized participants who are exposed to at least 1 dose of study intervention and have evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 100 | 86 | 110 | 87
percentage change | -50.68 (5.90) | -3.03 (7.07) | -58.72 (5.28) | -2.50 (6.95)
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model was used with baseline, geographic region, sex, treatment (Type III sum of squares) as covariates; LS Mean Change difference = -47.65, 95% CI 2-sided [-65.76 to -29.55]
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model was used with baseline, geographic region, sex, treatment (Type III sum of squares) as covariates; LS Mean Change difference = -56.21, 95% CI 2-sided [-73.73 to -38.70]

3. Secondary Outcome: Percentage of Participants With ≥50% AHI Reduction From Baseline
Description: Percentage of participants achieving ≥50% AHI reduction from baseline to Week 52 was evaluated.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 100 | 86 | 110 | 87
percentage of participants | 61.22 | 18.96 | 72.40 | 23.25
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 42.77, 95% CI 2-sided [30.76 to 54.79]
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 48.60, 95% CI 2-sided [36.55 to 60.65]

4. Secondary Outcome: Percentage of Participants With AHI <5 or With AHI 5-14 With Epworth Sleepiness Scale (ESS) ≤10
Description: The percentage of participants with OSA remission (AHI <5 events per hour of sleep) or with mild OSA without excessive daytime sleepiness (AHI 5-14 events per hour of sleep with ESS ≤10) at Week 52 was evaluated. The ESS is used to assess improvements in excessive daytime sleepiness from baseline to Week 52. The ESS is an 8-item, participant-completed measure that asks the participant to rate, on a scale of 0 (no chance of dozing) to 3 (high chance of dozing), their usual chances of dozing in 8 different daytime situations, with a recall period of "in recent times." The ESS total score is the sum of the 8-item scores and ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 100 | 86 | 110 | 87
percentage of participants | 42.17 | 15.88 | 50.24 | 14.33
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Test type: Superiority; p < .001, Regression, Logistic; Risk Difference (RD) = 28.74, 95% CI 2-sided [18.27 to 39.22]
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 33.22, 95% CI 2-sided [22.12 to 44.31]

5. Secondary Outcome: Change From Baseline in Sleep Apnea-Specific Hypoxic Burden (SASHB) (% Min/Hour)
Description: SASHB was determined by measuring the respiratory event-associated area under the curve for oxygen desaturation from pre-event baseline and represents the cumulative burden of intermittent hypoxia caused by OSA-related sleep-disordered breathing at sleep.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: %.min/hr
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 100 | 86 | 110 | 87
%.min/hr | -95.19 (4.081) | -25.07 (9.804) | -102.98 (3.758) | -41.69 (11.313)
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Test type: Superiority; Median Difference (Net) = -70.13, 95% CI 2-sided [-90.94 to -49.31], Standard Error of Mean 10.619
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Test type: Superiority; Median Difference (Net) = -61.29, 95% CI 2-sided [-84.66 to -37.93], Standard Error of Mean 11.921

6. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Sleep-Related Impairment 8a (PROMIS SRI) and PROMIS Short Form Sleep Disturbance 8b (PROMIS SD)
Description: PROMIS SRI consists of 8 items that assess self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours and perceived functional impairments associated with sleep problems. PROMIS SRI has a recall period of "in the past 7 days" and each item is rated on a 5-point scale from "not at all" to "very much." PROMIS SD consists of 8 items that assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. PROMIS SD has a recall period of "in the past 7 days" and each item is rated on a 5-point scale ranging from "not at all" to "very much," "never" to "always," or "very poor" to "very good." For both PROMIS SRI and PROMIS SD, item responses are used to generate T-scores which are standardized scores with a mean of 50 and a standard deviation of 10 (score range cannot be specified for T-scores). Higher T-scores indicate worse outcomes; more sleep-related impairment (PROMIS SRI) or more sleep disturbance (PROMIS SD).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: T score
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 90 | 79 | 93 | 79
T score
  Sleep Disturbance | -4.47 (0.69) | -2.44 (0.70) | -6.98 (0.82) | -3.08 (0.88)
  Sleep-Related Impairment: number analyzed (Participants) | 90 | 79 | 93 | 78
  Sleep-Related Impairment | -6.57 (0.83) | -3.13 (0.80) | -8.18 (0.95) | -3.91 (1.03)
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Sleep Disturbance; Test type: Superiority; p = 0.037, ANCOVA; ANCOVA model was used with baseline, geographic region, sex, baseline OSA severity Group, treatment (Type III sum of squares) as covariates; LS Mean Change difference = -2.03, 95% CI 2-sided [-3.95 to -0.12]
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Sleep Related Impairment; Test type: Superiority; p = 0.003, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Change difference = -3.43, 95% CI 2-sided [-5.69 to -1.17]
Statistical Analysis 3: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Sleep Disturbance; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Change difference = -3.90, 95% CI 2-sided [-6.21 to -1.58]
Statistical Analysis 4: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Sleep-Related Impairment; Test type: Superiority; p = 0.002, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Change difference = -4.26, 95% CI 2-sided [-6.97 to -1.56]

7. Secondary Outcome: Percent Change From Baseline in Body Weight
Description: Percent Change from Baseline in Body Weight was evaluated.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 101 | 87 | 113 | 90
Percent change | -17.65 (0.69) | -1.56 (0.68) | -19.62 (0.71) | -2.34 (0.74)
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Change difference = -16.09, 95% CI 2-sided [-17.99 to -14.19]
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Test type: Superiority; p < .001, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Change difference = -17.28, 95% CI 2-sided [-19.29 to -15.28]

8. Secondary Outcome: Change From Baseline in High Sensitivity C Reactive Protein (hsCRP) Concentration
Description: HsCRP is a marker for inflammation and was measured from blood samples to identify the presence of inflammation, to determine its severity, and to monitor response to treatment.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: Milligram per liter (mg/L)
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 95 | 84 | 102 | 82
Milligram per liter (mg/L) | -1.42 (0.151) | -0.70 (0.203) | -1.37 (0.130) | -0.33 (0.236)
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Test type: Superiority; p = 0.752, ANCOVA — ANCOVA model was used with baseline, geographic region, sex, baseline OSA severity Group, treatment (Type III sum of squares) as covariates; LS Mean Change difference = -0.71, 95% CI 2-sided [-1.21 to -0.22], Standard Error of Mean 0.253
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Test type: Superiority; p = 0.350, ANCOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean Change difference = -1.04, 95% CI 2-sided [-1.57 to -0.51], Standard Error of Mean 0.269

9. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Description: Change in systolic blood pressure from baseline to Week 48 was evaluated.
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mm Hg)
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
Number analyzed (Participants) | 100 | 89 | 112 | 91
Millimeters of mercury (mm Hg) | -9.46 (1.02) | -1.84 (1.03) | -7.64 (1.03) | -3.94 (1.18)
Statistical Analysis 1: Comparison: Tirzepatide MTD_GPI1 vs Placebo_GPI1; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Change difference = -7.62, 95% CI 2-sided [-10.48 to -4.77]
Statistical Analysis 2: Comparison: Tirzepatide MTD_GPI2 vs Placebo_GPI2; Test type: Superiority; p = 0.017, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean difference = -3.70, 95% CI 2-sided [-6.75 to -0.65]

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 56 Weeks)
Description: All randomized participants who are exposed to at least 1 dose of study intervention. As per the prespecified statistical analysis plan, adverse events were analyzed as per the treatment regimen. Gender-specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Tirzepatide MTD_GPI1 | Placebo_GPI1 | Tirzepatide MTD_GPI2 | Placebo_GPI2
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/120 | 0/119 | 0/114
Serious Adverse Events (participants affected / at risk) | 9/114 | 7/120 | 7/119 | 12/114
Other Adverse Events (participants affected / at risk) | 91/114 | 91/120 | 98/119 | 82/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tirzepatide MTD_GPI1 (N=114) | Placebo_GPI1 (N=120) | Tirzepatide MTD_GPI2 (N=119) | Placebo_GPI2 (N=114)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/78 (0) | 0/79 (0) | 0/87 (0) | 1/82 (1)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0/36 (0) | 0/41 (0) | 0/32 (0) | 1/32 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tirzepatide MTD_GPI1 (N=114) | Placebo_GPI1 (N=120) | Tirzepatide MTD_GPI2 (N=119) | Placebo_GPI2 (N=114)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Autoimmune thyroid disorder (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 5 (10) | 1 (1) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (4) | 5 (8) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 2 (6) | 7 (8) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon dysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 18 (25) | 3 (4) | 18 (19) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 30 (69) | 15 (21) | 26 (56) | 10 (15)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 2 (4) | 11 (11) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 9 (11) | 0 (0) | 10 (26) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (13) | 1 (1) | 6 (8) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malocclusion (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 29 (59) | 12 (15) | 26 (58) | 6 (7)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic floor dysfunction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 20 (34) | 5 (6) | 11 (18) | 1 (1)
Administration site reaction (General disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site reaction (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 4 (22) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (13) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 2 (13) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 8 (70) | 1 (2) | 6 (44) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Local reaction (General disorders) | 1 (2) | 0 (0) | 1 (8) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (4) | 2 (2) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 7 (7)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 6 (6) | 10 (11) | 8 (8) | 11 (12)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epstein-barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 4 (4) | 7 (8) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (5) | 8 (8) | 3 (3) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 8 (8) | 15 (24) | 12 (17)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 5 (5)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 10 (11) | 5 (7) | 8 (9)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 3 (5)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (2) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viiith nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Albumin urine present (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcitonin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 4 (5)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Blood osmolarity decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blood pressure measurement (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronavirus test positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine urine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 5 (5) | 2 (2) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 3 (4) | 0 (0) | 4 (5) | 0 (0)
Lipids abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sars-cov-2 test positive (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3) | 4 (4) | 0 (0) | 4 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 4 (4) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 2 (4) | 2 (2) | 1 (2) | 3 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 3 (6) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (3)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device physical property issue (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4) | 2 (2) | 2 (2) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rapid eye movement sleep behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 2 (2) | 3 (4) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/78 (0) | 0/79 (0) | 0/87 (0) | 1/82 (1)
Cervical cyst (Reproductive system and breast disorders) | 1/36 (1) | 0/41 (0) | 0/32 (0) | 0/32 (0)
Cervical polyp (Reproductive system and breast disorders) | 0/36 (0) | 0/41 (0) | 1/32 (1) | 0/32 (0)
Prostatitis (Reproductive system and breast disorders) | 1/78 (1) | 0/79 (0) | 0/87 (0) | 1/82 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/36 (0) | 1/41 (1) | 0/32 (0) | 0/32 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3) | 3 (3) | 2 (2)
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 5 (5) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cochlea implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fascia release (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 8 (9) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT05412004/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT05412004/SAP_001.pdf